CLINICAL TRIAL: NCT01648517
Title: Genotype-Driven Treatment of Advanced Non-small Cell Lung Cancer Based on mRNA Expression of ERCC1 & RRM1 as First-line Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2008-0132
Record Dates: First submitted 2012-07-01; First posted 2012-07-24 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Non-small Cell Lung Carcinoma
Keywords: on-small cell lung carcinoma; chemotherapy naive patient
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Genomic-driven dual agent chemotherapy Chemotherapy will consist of the assigned two drugs according to ERCC1 and RRM1 mRNA expression level A1: docetaxel + vinorelbine (DV) A2: gemcitabine + vinorelbine (GV) A3: docetaxel + carboplatin (DC) A4: gemcitabine + carboplatin (GC)
  Interventions: Drug: chemotherapy
- Arm B (Active Comparator): standard of care All control arm patients received standard platinum-based doublet chemotherapy with docetaxel plus carboplatin
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Drug: chemotherapy — A1: docetaxel 60mg/m2 on Day 1 vinorelbine 20mg/m2 on Day 1 and Day 8 (DV) A2: gemcitabine 1000mg/m2 on Day 1 vinorelbine 25mg/m2 on Day 1 and Day 8 (GV) A3: docetaxel 75mg/m2 on Day 1 carboplatin AUC5 on Day 1 (DC) A4: gemcitabine 1000mg/m2 on Day 1 and 8 carboplatin AUC5 on Day 1 (GC)
  Other Names: Docetaxel - Taxotere; Vinorelbine: Sandoz vinorelbine; Carboplatin: Carplan; Gemcitabine: Gemzar
  Arms: Arm A
Drug: chemotherapy — Drug: Docetaxel 75mg/m2 IV on Day 1 Drug: Carboplatin AUC5 IV on Day 1
  Other Names: Docetaxel - Taxotere; Carboplatin: Carplan
  Arms: Arm B

SUMMARY:
This is a prospective phase II trial, in patients with unresectable or metastatic NSCLC using chemotherapy regimens which will be defined according to the mRNA expression of ERCC1 and RRM1 of the tumor cells.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed unresectable advanced or metastatic non-small cell lung cancer (NSCLC) (stage IIIB or IV)
2. Chemotherapy naïve patient (Previous adjuvant or neoadjuvant chemotherapy allowed if the last dose was administered equal to or greater than 6 months ago.)
3. Age > 18
4. Performance status 0 to 2 by Eastern Cooperative Oncology Group (ECOG) criteria
5. At least one measurable lesion by Response Evaluation Criteria In Solid Tumors (RECIST)
6. Adequate organ functions (assessed within 14 days of starting treatment) 1) Bone marrow: Absolute neutrophil count ≥ 1,500/mm³, Platelet count ≥ 100,000/mm³, Hemoglobin ≥ 9.0 mg/dL 2) Liver: Total bilirubin ≤ 1.5 x ULN; aspartic transaminase (AST) and alanine transaminase (ALT), alkaline phosphatase(ALP) ≤ 2.5 x ULN 3) Kidney: Serum creatinine ≤ 1.5 x ULN
7. Signed informed consent document

Exclusion Criteria:

1. Clinically significant serious illness or medical condition (infection)
2. Prior systemic chemotherapy or immunotherapy for advanced NSCLC.
3. Presence of uncontrolled brain or leptomeningeal metastases
4. Prior radiotherapy within 3 weeks of starting treatment
5. Peripheral neuropathy equal to or greater than grade 2 by Common Terminology Criteria for Adverse Events (CTCAE) v4.0
6. Pregnant or lactating
7. Absolute contraindication of corticosteroid use
8. Patients with a history of severe hypersensitivity reaction to docetaxel, carboplatin, vinorelbine or gemcitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07-27 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
overall Response Rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  ORR was assessed by tumor response evaluation according to RECIST 1.1 at every 8 weeks. Tumor assessments will continue about every 8 weeks until disease progression or initiation of subsequent anticancer treatment.
  (If PR or CR was first documented, confirmation assessment was done between 4 weeks and 8 weeks)

SECONDARY OUTCOMES:
Progression free survival | up to 4 years
overall survival | up to 4 years
duration of response | up to 4 years
disease control rate | up to 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Heo SJ, Jung I, Lee CK, Kim JH, Lim SM, Moon YW, Shim HS, Jeong J, Kim JH, Kim HR, Cho BC. A randomized phase II trial of ERCC1 and RRM1 mRNA expression-based chemotherapy versus docetaxel/carboplatin in advanced non-small cell lung cancer. Cancer Chemother Pharmacol. 2016 Mar;77(3):539-48. doi: 10.1007/s00280-016-2968-z. Epub 2016 Jan 25. PMID 26811178